CLINICAL TRIAL: NCT06373003
Title: Negative Antiphospholipid Syndrome: a Multicentric Study
Status: Recruiting | Type: Observational
Sponsor: Italian Society for Rheumatology (Other)
Responsible Party: Sponsor
Other Study IDs: SNAPSITA
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Antiphospholipid Syndrome; Seronegative Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected on two occasions at least 12 weeks apart for each patient; the aPL criteria will be tested in each recruitment centre, as a routine practice, whilst the non-criterion aPL will be tested in the centralized laboratory at the Department of "Experimental Medicine', Umberto I Polyclinic in Rome
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 [APS]: Patients fulfilling the classification criteria for antiphospholipid syndrome (seropositive APS, SN-APS)
  Interventions: Other: Diagnostic accuracy
- Group 2 [SN-APS]: Patients with seronegative APS (SN-APS): with clinical criteria (thrombotic or obstetric) for APS, persistently negative for aPL, and with clinical features highly suggestive of APS (recurrent events, thrombotic + obstetrical events, extra-criteria manifestations, other autoimmune diseases)
  Interventions: Other: Diagnostic accuracy
- Group 3 [Control Group]: Patients with clinical criteria (thrombotic or obstetric) for APS, negative for aPL, but without clinical features highly suggestive of APS (recurrent events, thrombotic + obstetrical events, extra-criteria manifestations, other autoimmune diseases)

INTERVENTIONS:
Other: Diagnostic accuracy — To assess the diagnostic accuracy of non-criteria aPL (anti-vimentin/cardiolipin and anti-phosphatidylserine/prothrombin) in identifying APS in patients with thrombosis/ recurrent adverse pregnancy outcomes
  Groups: Group 1 [APS]; Group 2 [SN-APS]

SUMMARY:
Multicentre no-profit, national, (cross-sectional diagnostic) retrospective study, promoted by the Italian Society for Rheumatology.

The main objective of the study is to assess the diagnostic accuracy of non-criteria aPL (anti-vimentin/cardiolipin and anti-phosphatidylserine/prothrombin) in identifying APS in patients with thrombosis/recurrent adverse pregnancy outcomes.

DETAILED DESCRIPTION:
BACKGROUND Antiphospholipid syndrome (APS) is an autoimmune disorder leading to arterial and/or venous thrombotic events, and pregnancy morbidity. Seronegative antiphospholipid syndrome (SN-APS) occurs in case of clinical manifestations highly suggestive of APS but with negative test for circulating conventional antiphospholipid antibodies (anticardiolipin antibodies, anti-beta-I-glycoprotein antibodies, lupus anticoagulant). Recent studies have shown that most SN-APS patients present circulating (non-criteria) antibodies potentially explaining the clinical manifestations. In a smaller proportion of SN-APS patients, no antibody has been detected so far. Available knowledge on the clinical presentation and disease course of SN-APS is limited, and the causal relationship between non-criteria antibodies and recurrent thrombosis deserves further research to be confirmed. To date, no difference between APS and SN-APS groups has been highlighted in terms of thrombotic events or pregnancy morbidity, but this could be in part explained by small samples not sufficiently powered to detect a difference. Moreover, it is still to determine whether the detection of "non-criteria" antibodies in addition to conventional aPL may help stratify patients according to their risk of clinical manifestation.A multicentre study involving Italian centres could allow to investigate the diagnostic accuracy of no-criteria aPL and elucidate the prognostic impact of such antibodies alone or in combination with criteria aPL. In addition, a multicentre study could allow to study a larger sample of patients and better quantify poorly investigated aspects in SN-APS

MAIN OBJECTIVE To assess the diagnostic accuracy of non-criteria aPL (anti-vimentin/cardiolipin and anti-phosphatidylserine/prothrombin) in identifying APS in patients with thrombosis/recurrent adverse pregnancy outcomes (group 1 vs group 3, see below).

SECONDARY OBJECTIVES

* To assess the diagnostic accuracy of non-criteria aPL in identifying SN-APS in patients with thrombosis/recurrent adverse pregnancy outcomes (group 2 vs group 3).
* To compare the clinical characteristics of APS vs SN-APS in patients with and without non-criteria aPL.
* To estimate the association between different aPL status on the recurrence of thrombosis/adverse pregnancy outcomes.

EXPLORATORY OBJECTIVE To assess the prevalence of: anti-cardiolipin antibodies (aCL) by thin-layer chromatography (TLC)-immunostaining, anti-carbamylated-β2-glycoprotein I antibodies and Anti-glucose-modified β2 glycoprotein I antibodies in APS and SN-APS groups (group 1 and group 2).

SAMPLE SIZE AND STUDY PROCEDURES A minimum sample size of 35 patients for each group is planned for this study

LABORATORY PROCEDURES Blood samples will be collected and analysed in each recruiting centre, as routine practice at 12 weeks apart. The laboratory tests for the non-criteria aPL will be centrally performed at the Department of "Experimental Medicine', Umberto I Polyclinic in Rome.

STUDY DURATION Enrolment: 24 months starting from the first patient recruited Analysis and reporting: 12 months starting from the end of the enrollment

STUDY SCHEME The study can be divided into three phases: i) the collection of all clinical data at the onset of the thrombotic or obstetric event; ii) the collection of all the clinical data between the first clinical event and the patient recruitment; iii) the detection of non-criteria aPL from the patient's blood samples. The first two phases characterise the retrospective part of the study, while the third phase characterises the cross-sectional part of the study.

In phase 1, the following data associated with the clinical event will be collected: relevant demographic data, the history of all criteria events, the history of all non-criteria events, all relevant risk factors, the history of pharmacological treatments before or in progress at the clinical event and the collection of laboratory data available at the diagnosis. Phase 1 data will be collected by all participating centres.

In phase 2, new criteria events, non-criteria manifestations related to the clinical events and risk factors developed between the first clinical event and the date of recruitment of a patient will be assessed. Phase 2 data will be collected by all participating centres.

In phase 3, patients' blood samples will be tested at the coordinating centre to evaluate the presence of non-criteria aPL. Two blood samples will be collected by each patient recruited by a centre; such samples should be primarily retrieved from those previously collected by a centre at the time of diagnosis(herein "serum library") and stored at the centre itself; in case of their absence, blood samples can be collected from a recruited patient upon enrolment. In case only one sample can be retrieved from the hospital serum library, the remaining one will be collected from the recruited patient. Blood samples taken from deceased patients will be excluded.

STATISTICAL ANALYSIS Baseline characteristics will be summarized by descriptive statistics. The accuracy of non-criteria aPL (index test) in discriminating between cases and controls (reference standard) will be estimated as sensitivity and specificity.

A first analysis will use APS criteria cases (group 1) and controls(group 3) as non-cases; a second analysis will use SN-APS (group 2) as cases and controls (group 3) as non-cases.

The following groups [APS (group 1), SN-APS (group 2 subdivided into positive for non-criteria aPL and negative for non-criteria) and controls (group 3)] will be compared for clinical characteristics treatment variables.

A logistic regression model, considering the recurrent event as outcome and the APS status (groups 1, 2 and 3) as predictor, adjusted for demographic, event type and treatment will be performed

ELIGIBILITY:
INCLUSION CRITERIA:

1. Group 1 [APS]: Patients fulfilling the classification criteria for antiphospholipid syndrome (seropositive APS, SP-APS)
2. Group 2 [SN-APS]: patients with seronegative APS (SN-APS): with clinical criteria (thrombotic or obstetric) for APS, persistently negative for aPL, and with clinical features highly suggestive of APS (recurrent events, thrombotic + obstetrical events, extra-criteria manifestations, other autoimmune diseases)
3. Group 3: patients with clinical criteria (thrombotic or obstetric) for APS, negative for aPL, but without clinical features highly suggestive of APS (recurrent events, thrombotic + obstetrical events, extra-criteria manifestations, other autoimmune diseases).
4. Age < 65 years (at event time)
5. Less than 5 years from the first even

EXCLUSION CRITERIA

1. Group 2 and 3: patients with a known cause of thrombosis or obstetrical manifestations
2. Deceased patients
3. Less than 5 years from the first event

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators plan to include a minimum sample size of 35 patients for each group; all patients will have the following features:
  * patients affected by Antiphospholipid syndrome (APS) or Seronegative antiphospholipid syndrome (SN-APS) or patients with clinical criteria (thrombotic or obstetric) for APS, negative for aPL, but without clinical features highly suggestive of APS
  * Age <65 years (at the event time)
  * Less than 5 years from the first event to the beginning of the study
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2024-09-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of non-criteria aPL | 0 months
  Evaluation of the sensitivity and specificity of non-criteria aPL (anti-vimentin/cardiolipin and anti-phosphatidylserine/prothrombin) in identifying APS in patients with thrombosis/recurrent adverse pregnancy outcomes

SECONDARY OUTCOMES:
Frequency of clinical characteristics in the aPL groups | 0 months
  Assessment of the frequency of clinical characteristics in the four different aPL status groups, including APS and SN-APS with and without non-criteria aPL
Incidence of recurrent thrombosis and pregnancy complications | 0 months
  Aestimation of the association between different aPL status on the recurrence of thrombosis/adverse pregnancy outcomes.

OTHER OUTCOMES:
Prevalence of APS- and SN-APS-related antibodies in study groups | 0 months
  Prevalence of aCL by TLC-immunostaining, anti-carbamylated-β2-glycoprotein I antibodies and Anti-glucose-modified β2 glycoprotein I antibodies in APS and SN-APS groups

CONTACTS AND LOCATIONS:
Locations (1):
- Umberto I Polyclinic, Rome- Department of Rheumatology, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
The Italian Society of Rheumatology (SIR) is the only data controller of the study and only reports containing aggregated analysed data will be shared.